CLINICAL TRIAL: NCT01013454
Title: A Phase 1, Open-Label, Single Dose Study To Characterize The Pharmacokinetics Of A Varenicline (CP-526,555) Transdermal Delivery System Applied To The Skin Of Adult Smokers
Brief Title: A Study Evaluating The Absorption Of Varenicline Into The Body From A Varenicline Patch Applied To The Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3051119
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Smoking Cessation
Keywords: varenicline percutaneous transcutaneous topical transdermal transdermal delivery system patch
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varenicline transdermal delivery system (Experimental)
  Interventions: Drug: varenicline free base patch

INTERVENTIONS:
Drug: varenicline free base patch — varenicline transdermal delivery system (6.0 mg payload [drug amount loaded in each patch]) will be applied to the upper back over a single 24 hour period

SUMMARY:
This study will evaluate the single-dose pharmacokinetics, safety, and tolerability of a varenicline patch applied to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Caucasian, male, adult light to regular smokers

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption through the skin (eg, psoriasis).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Varenicline area under the curve from 0 to infinity (AUCinf) and varenicline area under the curve from 0 to the last quantifiable concentration (AUClast), as data permit | 8 days

SECONDARY OUTCOMES:
Evaluation of adverse events (including skin irritation) | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051119&StudyName=A%20Study%20Evaluating%20The%20Absorption%20Of%20Varenicline%20Into%20The%20Body%20From%20A%20Varenicline%20Patch%20Applied%20To%20The%20Skin